CLINICAL TRIAL: NCT04599244
Title: Assessment of the Effect of Emergency Pulpotomy Versus Complete Pulp Extirpation on Anesthetic Efficacy in Endodontic Treatment of Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Effect of Emergency Pulpotomy Versus Pulp Extirpation on Anesthetic Efficacy in Endodontic Treatment of Acute Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Ali, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3-3-5
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Symptomatic Irreversible Pulpits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- emergency pulpotomy (Experimental): intervention arm
  Interventions: Other: emergency pulpotomy
- complete pulp extirpation (Active Comparator): control arm
  Interventions: Other: emergency pulpotomy

INTERVENTIONS:
Other: emergency pulpotomy — removal of coronal pulp

SUMMARY:
Irreversible pulpitis is an inflammatory condition of the dental pulp, highly painful, and one of the main reasons for seeking emergency dental treatment. Pain associated with irreversible pulpitis represents more than 45% of emergency patients in dental clinics. A pulpotomy has been demonstrated as an emergency intervention for effective pain relief by removing the coronal pulp tissue without penetrating radicular pulpal tissue. Inflammation and degeneration of the pulp usually progress apically from the point of infection, so selective removal of this tissue in the form of pulpotomy is usually effective in controlling pain and patient sedation.

The rationale behind emergency pulpotomy is relieving acute dental pain caused by irreversible pulpitis. However, there is still insufficient evidence to determine whether the presence, nature and duration of clinical symptoms gives accurate information about the extent of pulp inflammation, as pulpotomy was found to be an effective emergency treatment strategy with respect to relieving clinical symptoms, even in cases of irreversible pulpitis with symptomatic apical periodontitis . Advanced diagnostic strategies are needed to determine whether there is a correlation between clinical symptoms, actual pulpal inflammation and achieving adequate pain relief during and after treatment. Thus, we are conducting this study to assess the effect of emergency pulpotomy versus complete pulp extirpation on relieving acute dental pain of symptomatic irreversible pulpitis in mandibular molars. The expected benefit for the patients is to decrease pain during and after treatment. we also are trying to provide an evidence for the clinician in order to provide the best endodontic treatment without pain.

DETAILED DESCRIPTION:
Irreversible pulpitis is an inflammatory condition of the dental pulp, highly painful, and one of the main reasons for seeking emergency dental treatment. Pain associated with irreversible pulpitis represents more than 45% of emergency patients in dental clinics. A pulpotomy has been demonstrated as an emergency intervention for effective pain relief by removing the coronal pulp tissue without penetrating radicular pulpal tissue. Inflammation and degeneration of the pulp usually progress apically from the point of infection, so selective removal of this tissue in the form of pulpotomy is usually effective in controlling pain and patient sedation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are medically free from any systemic disease that may contra indicate our interventions.
* Patient's age between 18-65 years old.
* Mandibular molar having vital pulps with symptomatic irreversible pulpitis because this group of patients may have more endodontic pain
* Positive patient's acceptance for participation in the study.

Exclusion Criteria:

* - Patients who had used any type of analgesic medication during the preceding 12 hours before the treatment to give true response of pain during treatment.
* Teeth with necrotic pulp.
* Pregnant patients or lactating because of radiographic hazards and use of analgesics.
* Any known sensitivity or adverse reactions to ibuprofen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
anesthetic efficacy | During pulp extirpation and pulpotomy (30 minutes)
  measured byVerbal rating scale (VRS),unit:Binary (success/failure)

IPD SHARING:
Plan to Share IPD: Undecided